CLINICAL TRIAL: NCT00084682
Title: A Phase II Study of Single Agent Depsipeptide (FK228; NSC 630176; IND 51,810) in Patients With Unresectable Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Depsipeptide in Unresectable Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00027; MMC 04-02-025S (Other: Montefiore Medical Center); N01CM62204 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (romidepsin) (Experimental): Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax

SUMMARY:
This phase II trial is studying how well FR901228 works in treating patients with unresectable recurrent or metastatic squamous cell carcinoma (cancer) of the head and neck. Drugs used in chemotherapy such as FR901228 work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the rate of disease control (i.e., achievement of complete response, partial response, or stable disease) of the single agent depsipeptide in patients with unresectable recurrent or metastatic squamous cell carcinoma of the head and neck.

SECONDARY OBJECTIVES:

I. To evaluate the duration of response, time to progression, and overall survival for patients with incurable head and neck cancer treated with depsipeptide.

TERTIARY OBJECTIVES:

I. To determine the extent of histone hyperacetylation in peripheral blood mononuclear cells (PBMCs) as a readout of depsipeptide activity before and after depsipeptide administration, to correlate this activity with observed histone hyperacetylation in tumor and mucosal cells, and to correlate extent of depsipeptide activity with tumor response.

II. To determine depsipeptide-induced changes in the gene expression profile of tumor cells from biopsies of accessible tumor tissue and of mucosal cells from transepithelial oral brush biopsies using cDNA microarrays containing 28,000 clones, and to correlate these changes with extent of histone hyperacetylation observed in PBMCs and tumor tissues.

III. To determine depsipeptide-induced changes in methylation of candidate genes in tumor cells and oral mucosa epithelia.

IV. To demonstrate altered expression of signaling and cell cycle-related proteins in tumor tissue in response to depsipeptide.

OUTLINE: This is a multicenter study.

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed squamous cell cancer of the head and neck (MedDRA code 90002024), excluding nasopharyngeal primaries, which is unresectable or metastatic; the disease must be incurable with surgery or radiation therapy; the tumor should preferably be present at the primary site, and it must be accessible to planned biopsy methods
* Measurable disease by RECIST,
* May have received any number of prior systemic chemotherapy regimen for unresectable, recurrent or metastatic disease; if the only site of measurable disease is a previously irradiated area, the patient must have documented progressive disease or biopsy-proven residual carcinoma; persistent disease after radiotherapy must be biopsy-proven at least 8 weeks after the completion of radiotherapy
* Life expectancy of greater than 3 months
* Normal organ and marrow function as defined by the following labs performed =< 2 weeks of study entry:
* Leukocytes ≥ 3,000/uL
* Absolute Neutrophil Count ≥ 1,500/uL
* Hemoglobin ≥ 10 gm%
* Platelets ≥ 100,000/uL
* Total Bilirubin =< 1.5 X upper normal institutional limit
* AST(SGOT)/ALT(SGPT) =< 2.5 X upper normal institutional limits
* Creatinine within normal institutional limits OR creatinine clearance ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* PT/PTT =< 1.1X upper normal institutional limits
* Calcium within normal institutional limits
* CPK, Troponin within normal institutional limits
* Uric Acid within normal institutional limits
* Ability to understand and the willingness to sign a written informed consent document; in addition to consent for the therapy, patients must give consent to required pre- and post-therapy blood and tissue samples;

Exclusion Criteria:

* Patients should not have had prior therapy with depsipeptide and may not be receiving any other investigational agents or drugs known to have histone deacetylase inhibitor activity such as sodium valproate
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Significant cardiac disease including congestive heart failure that meets New York Heart Association (NYHA) class III and IV definitions (see Appendix II), history of myocardial infarction within one year of study entry, uncontrolled dysrhythmias, or poorly controlled angina
* History of serious ventricular arrhythmia (VT or VF, > 3 beats in a row), QTc > 500 msec, or LVEF < 40%
* Patients may not be co-medicated with an agent that causes QTc prolongation; - Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Not pregnant or lactating
* History of HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-06; Primary Completion 2008-11 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Missak Haigentz, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Result] Haigentz M Jr, Kim M, Sarta C, Lin J, Keresztes RS, Culliney B, Gaba AG, Smith RV, Shapiro GI, Chirieac LR, Mariadason JM, Belbin TJ, Greally JM, Wright JJ, Haddad RI. Phase II trial of the histone deacetylase inhibitor romidepsin in patients with recurrent/metastatic head and neck cancer. Oral Oncol. 2012 Dec;48(12):1281-8. doi: 10.1016/j.oraloncology.2012.05.024. Epub 2012 Jun 28. PMID 22748449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 patients were enrolled from one institution between June 2005 and October 2008
Groups:
- Treatment (Romidepsin): Patients receive FR901228 (depsipeptide) IV at 13 mg/m2 over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  romidepsin: Given IV
Period: Overall Study
Arm/Group | Treatment (Romidepsin)
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Romidepsin)
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 59.0 [46 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7
  Black | 1
  Hispanic | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease Control (i.e., Achievement of Complete Response, Partial Response, or Stable Disease)
Description: Tumor response was assessed every eight weeks per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions as assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Stable disease (SD) was defined as having no evidence of response (CR or PR) as best response to therapy, and no evidence of disease progression (appearance of new lesions or >/= 30% increase in target lesions) at 8 weeks.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Treatment (Romidepsin): Patients receive FR901228 (depsipeptide) IV at 13 mg/m^2 over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  romidepsin: Given IV
Arm/Group | Treatment (Romidepsin)
Number analyzed (Participants) | 13
participants
  Stable Disease | 2 [1.9 to 45.5]
  Disease progression | 9 [1.9 to 45.5]
  Symptomatic deterioration | 2 [1.9 to 45.5]

2. Secondary Outcome: Duration of Response
Time Frame: Up to 2 years
Population: Data not collected. As the first stage goal of 8 patients with disease control was not achievable, further analysis was not done.
Arm/Group | Treatment (Romidepsin)
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Progression
Description: All time to event endpoints will be evaluated using Kaplan Meier estimates and survival curves will be generated based on these estimates.
Time Frame: Up to 2 years
Population: Data not collected. As the first stage goal of 8 patients with disease control was not achievable, further follow up was not done.
Arm/Group | Treatment (Romidepsin)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: All time to event endpoints will be evaluated using Kaplan Meier estimates and survival curves will be generated based on these estimates. One and two-year survival and median survival time (if attained) will be estimated and reported with 95% confidence limits. If the sample sizes are sufficient, subgroup analysis based on baseline factors will be performed using the log rank test to compare survival curves.
Time Frame: Up to 2 years
Population: data not collected
Arm/Group | Treatment (Romidepsin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Romidepsin)
Serious Adverse Events (participants affected / at risk) | 12/14
Other Adverse Events (participants affected / at risk) | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Romidepsin) (N=14)
Anemia (Blood and lymphatic system disorders) | 2 (14)
Thrombocytopenia (Investigations) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Lung infection (Infections and infestations) | 3 (3)
Soft tissue infection (Infections and infestations) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Romidepsin) (N=14)
Hypertension (Vascular disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less